CLINICAL TRIAL: NCT01872780
Title: The Effect of CYP2C8 E274Q, a Novel 23452 G>T SNP, on the Disposition of Rosiglitazone in Healthy Subjects: The Genetic Polymorphisms of CYP2C8 in a Korean Population
Brief Title: Identification of Null Allelic Variant of CYP2C8 In A Korean Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Department of Pharmacology and Pharmacogenomics Research Center, Inje University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08-101
Record Dates: First submitted 2011-12-06; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: CYP2C8; genetic polymorphism; rosiglitazone; Korean
MeSH Terms: interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rosiglitazone (Active Comparator): avandia
  Interventions: Drug: Rosiglitazone; Genetic: CYP2C8 genotype
- genetic polymorphism (Active Comparator): avandia CYP2C8 genotype
  Interventions: Drug: Rosiglitazone; Genetic: CYP2C8 genotype

INTERVENTIONS:
Drug: Rosiglitazone — single oral administration of 4mg of rosiglitazone
  Other Names: Avandia
Genetic: CYP2C8 genotype — CYP2C8*11.
  Other Names: avandia

SUMMARY:
The genotype profile of CYP2C8 was analyzed in a Korean population. Frequency in multi-ethnic population and in vivo functionality of novel null allelic CYP2C8 variant were evaluated.

DETAILED DESCRIPTION:
Whole blood samples from 50 unrelated Korean subjects were genotyped for 3kb of 5' upstream region, all exon-intron boundaries, exons, and UTR regions of CYP2C8 gene by direct sequencing. Genotyping of CYP2C8 has been addressed only for null allelic variant, CYP2C8*11 using pyrosequencing in the 447 Koreans, 93 African-Americans, 100 Caucasians, 348 Chineses and 100 Vietnameses. Then, in-vivo single PK study of CYP2C8 probe, rosiglitazone(4mg), was conducted in 7 healthy subjects with CYP2C8*1/*1 and 2 with CY2C8*1/*11.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Exclusion Criteria:

* Medical problems in taking probe drug

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
AUC | 12hr
  0h,0.33h,0.66h,1h,1.5h,2h,3h,4h,6h,8h,12h,24h

SECONDARY OUTCOMES:
Cmax | 12hr
  0h,0.33h,0.66h,1h,1.5h,2h,3h,4h,6h,8h,12h,24h

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, MD, PhD, Principal Investigator — Inje University